CLINICAL TRIAL: NCT04747821
Title: A Stepped-wedge Cluster Randomized Trial to Assess the Effectiveness of the Use of the Adsorbed COVID-19 (Inactivated) Vaccine Manufactured by Sinovac
Brief Title: An Effectiveness Study of the Sinovac's Adsorbed COVID-19 (Inactivated) Vaccine
Acronym: ProjetoS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COV-04-IB
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-02

CONDITIONS: Covid19
Keywords: COVID-19 Vaccines; Vaccines, Inactivated
MeSH Terms: conditions — COVID-19 | interventions — Vaccines; sinovac COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Groups of cluster are allocated to offer vaccination in a stepped-wedge mode.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First group of clusters (Experimental): Adsorbed COVID-19 (Inactivated) vaccine offered in the first week of study The vaccine is administrated in two doses with a four-weeks interval
  Interventions: Biological: Adsorbed COVID-19 (Inactivated) Vaccine
- Second group of clusters (Experimental): Adsorbed COVID-19 (Inactivated) vaccine offered in the second week of study The vaccine is administrated in two doses with a four-weeks interval
  Interventions: Biological: Adsorbed COVID-19 (Inactivated) Vaccine
- Third group of clusters (Experimental): Adsorbed COVID-19 (Inactivated) vaccine offered in the third week of study The vaccine is administrated in two doses with a four-weeks interval
  Interventions: Biological: Adsorbed COVID-19 (Inactivated) Vaccine
- Fourth group of clusters (Experimental): Adsorbed COVID-19 (Inactivated) vaccine offered in the fourth week of study The vaccine is administrated in two doses with a four-weeks interval
  Interventions: Biological: Adsorbed COVID-19 (Inactivated) Vaccine

INTERVENTIONS:
Biological: Adsorbed COVID-19 (Inactivated) Vaccine — Adsorbed COVID-19 (inactivated) Vaccine manufactured by Sinovac
  Other Names: CoronaVac

SUMMARY:
This is a stepped-wedge cluster randomized trial to assess effectiveness of Sinovac's Adsorbed COVID-19 (Inactivated) vaccine. Residents in the urban area of a municipality are eligible to participate. The city was divided in clusters and those cluster were grouped to determine the offer of vaccination in four steps. The vaccine will be offered to adults (18 years old and above) according to the location of their homes in a cluster. The vaccine schedule is two doses with four-weeks interval. Baseline samples to determine previous immunity will be collected before vaccination.

Cases of COVID-19 reported in the city will be recorded according to the WHO clinical progression scale. Comparison of periods before and after vaccination and relation to immunization coverage will be considered for the assessment of effectiveness in the clusters and groups of clusters.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age or older;
2. Resident in the study area;
3. Show voluntary intention to participate in the study, documented by the informed consent form signed by participant.

Exclusion Criteria:

1. For females: Pregnancy (confirmed by positive beta-hCG test), breastfeeding or intent to engage in sexual relations with reproductive intent without use of birth control methods in the three months following vaccination;
2. Evidence of uncontrolled neurological, cardiac, pulmonary, hepatic or renal disease, according to anamnesis or physical examination. Significant changes in treatment or hospitalizations due to worsening of the condition in the last three months are indicators of uncontrolled disease;
3. Diseases with impaired immune system including: neoplasms (except basal cell carcinoma), congenital or acquired immunodeficiencies and autoimmune diseases not controlled according to anamnesis or physical examination. Significant changes in treatment or hospitalizations due to worsening of the condition in the last three months are indicators of uncontrolled disease;
4. Behavioral, cognitive or psychiatric disease that, in the opinion of the principal investigator or his or her representative physician, affects the participant's ability to understand and cooperate with all study protocol requirements;
5. Any alcohol or drug abuse over the 12 months prior to enrollment in the study that has caused medical, professional or family problems, indicated by clinical history;
6. History of severe allergic reactions or anaphylaxis to the study vaccine or to components thereof;
7. History of asplenia;
8. Participation in another clinical trial with an investigational product in the six months prior to enrollment in the study or planned participation in another clinical trial within the two years following enrollment;
9. Previous participation in a study to evaluate a COVID-19 vaccine or prior exposure to a COVID-19 vaccine;
10. Use of immunosuppressant therapy regimens within the six months prior to enrollment in the study for planned use within the two years following enrollment. Immunosuppressant therapy regimens include: antineoplastic chemotherapy, radiation therapy and immunosuppressants to induce transplant tolerance, among others.
11. Use of immunosuppressive doses of corticosteroids within the three months prior to the enrollment in the study and planned use of immunosuppressive doses of corticoids within the three months following enrollment in the study. Immunosuppressive doses of corticosteroids will be considered the equivalent prednisone 20 mg/day for adults, for longer than one week. Continued use of topical or nasal corticosteroids is not considered an immunosuppressant;
12. Received blood products (transfusions or immunoglobulins) within the three months prior to enrollment in the study, or planned administration of blood products or immunoglobulins within the two years following enrollment in the study;
13. Suspected or confirmed fever within the 72 hours prior to vaccination or axillary temperature greater than 37.8 °C* on the day of vaccination (enrollment may be postponed until participant has gone 72 hours without fever);
14. Possible or confirmed case of COVID-19 on the day of vaccination (vaccination can be postponed until the participant completes 72 hours without symptoms or the diagnosis is ruled out);
15. Received live attenuated virus vaccine or inactivated vaccine within the 28 days or 14 days, respectively, prior to enrollment in the study, or immunization planned within the 28 days after enrollment in the study;
16. History of bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture
17. Any other condition that, in the opinion of the principal investigator or his/her representative physician, could put the safety/rights of potential participants at risk or prevent them from complying with this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27711 (Actual)
Dates: Start 2021-02-07 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of COVID-19 cases after two-doses immunization schedule in clusters in the first quarter of study | Thirteen weeks after the beginning of study vaccination
  Number of virologically-confirmed symptomatic COVID-19 six weeks after beginning of study vaccination up to thirteen weeks

SECONDARY OUTCOMES:
Incidence of COVID-19 cases after two-doses immunization schedule in clusters up to one year of study | One year after the beginning of study vaccination
  Number of virologically-confirmed symptomatic COVID-19 six weeks after beginning of study vaccination up to one year
Incidence of COVID-19 cases after two-doses immunization schedule in clusters according to immunization status | One year after the beginning of study vaccination
  Number of virologically-confirmed symptomatic COVID-19 six weeks after beginning of study vaccination up to one year according to immunization status
Incidence of COVID-19 cases after two-doses immunization schedule in clusters according to pre-existing SARS-CoV-2 antibodies | One year after the beginning of study vaccination
  Number of virologically-confirmed symptomatic COVID-19 six weeks after beginning of study vaccination up to one year according to pre-existing SARS-CoV-2 antibodies
Incidence of COVID-19 cases after two-doses immunization schedule in clusters according to immunization coverage | One year after the beginning of study vaccination
  Number of virologically-confirmed symptomatic COVID-19 six weeks after beginning of study vaccination up to one year according to immunization coverage
Incidence of hospitalization and death due to COVID-19 after two-doses immunization schedule in clusters | One year after the beginning of study vaccination
  Number of hospitalization and death due to COVID-19 six weeks after beginning of study vaccination up to one year
Change in average number of reported COVID-19 cases in the study area in comparison to other neighboring cities | One year after the beginning of study vaccination
  Average number of reported COVID-19 cases in the microregion where the study area is located
Medically-attended adverse reactions to the study vaccine | One week after each vaccination
  Number of medically-attended adverse reactions to the study vaccine
Frequency of severe COVID-19 cases | From first vaccination up to one year after first dose
  Frequency of virologically-confirmed severe COVID-19 cases after receiving, at least, one dose of the vaccine
Frequency of adverse events of special interest after immunization | From first vaccination up to one year after first dose
  Frequency of adverse events of special interest after receiving, at least, one dose of the vaccine
Acceptability of the study vaccine | Two weeks after the beginning of study vaccination of the corresponding cluster
  Acceptability rate of the study vaccine in the eligible population of each cluster
Adherence to vaccination schedule | Six weeks after the beginning of study vaccination of the corresponding cluster
  Adherence rate to vaccination schedule in the population of each cluster

OTHER OUTCOMES:
Frequency of SARS-CoV-2 variants in the study area | One year after the beginning of study vaccination
  Description of SARS-CoV-2 variants sequenced out of the samples collected in the study area

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Boulos, MD, MSc, Study Director — Butantan Institute
Locations (1):
- Hospital Estadual de Serrana, Serrana, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided